CLINICAL TRIAL: NCT05080140
Title: Investigate the Effect of Ezetimibe, Simvastatin, and Omega 3- Fatty Acids on Dyslipidemia Patients: a Pharmacokinetics Based Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Yasmine Farouk, Teacher Assistant - clinical pharmacy department, Misr University for Science and Technology
Other Study IDs: 1606YAS141008
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hyperlipidemia; Mixed
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Simvastatin
- Ezetimibe
  Interventions: Drug: Ezetimibe 10mg
- Omega -3 fatty acids-
- Simvastatin+ Ezetimibe
  Interventions: Drug: Ezetimibe 10mg
- Simvastain + ezetimibe + omega
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Ezetimibe 10mg — Effect of ezetimibe on hyperlipidemia on patients with diabetes mellites
  Groups: Ezetimibe; Simvastain + ezetimibe + omega; Simvastatin+ Ezetimibe

SUMMARY:
This randomized controlled pharmacokinetic based study will be carried out on patients with both sexes and various ages, plasma triglycerides levels, clinical health disorders and using different agents for treatment of their hyperlipidemia in order to access the optimal drug therapy with best cost effectiveness in the elderly cases under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of dyslipidemia with high triglyceride level (200 to 499 mg/100 ml).
* Total cholesterol level more than 200 mg/100 ml
* Male and female
* Age 35 - 70 years

Exclusion Criteria:

* - Hypersensitivity of drugs
* Liver toxicity
* -Patients suffering from renal dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: least 80 adult patients both sexes suffering from mixed dyslipidemia with high triglyceride level admitted at Sauad Kaffafi Hospital, Misr University for science and technology.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Reduction of Total cholesterol | 3 months
  reduction of LDL

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University for science and technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
result and conclusion sharing